CLINICAL TRIAL: NCT02394626
Title: RESURGE - Randomized Controlled Comparative Phase II Trial on Surgery for Glioblastoma Recurrence
Brief Title: Surgery for Recurrent Glioblastoma
Acronym: RESURGE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 368/14
Record Dates: First submitted 2015-03-11; First posted 2015-03-20 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
Keywords: Recurrent glioblastoma; Surgery; Complete resection of enhancing tumor; Survival; Quality of life
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery followed by adjuvant second-line therapy (Experimental): Surgery followed by adjuvant second-line therapy
  Interventions: Procedure: Surgery followed by adjuvant second-line therapy
- Second-line therapy alone (Active Comparator): Second-line therapy alone
  Interventions: Procedure: Second-line therapy alone

INTERVENTIONS:
Procedure: Surgery followed by adjuvant second-line therapy — Surgery:
  Surgery must take place between day 1 and 14 after study inclusion and within 21 days from the MRI on which recurrence was diagnosed. The modalities of surgery and the choice of pre- and intra-operative technical adjuncts is at the treating neurosurgery discretion. Surgery must take place between day 1 and 14 after study inclusion and within 21 days from the MRI on which recurrence was diagnosed. The modalities of surgery and the choice of pre- and intra-operative technical adjuncts is at the treating neurosurgery discretion. However, some form of intra-operative resection control (iMRI or intra-operative fluorescence) and function control (electrophysiology) should be available to the surgeon and used when warranted.
  Adjuvant second-line therapy:
  Patients will be seen after surgery by the treating neurooncologist. Modalities of adjuvant second-line therapy are individually defined according to local guidelines and are not stipulated by study protocol.
  Arms: Surgery followed by adjuvant second-line therapy
Procedure: Second-line therapy alone — Patients randomized to the non-surgical cohort receive second-line therapy according to local guidelines. Modalities thereof are not stipulated by study protocol.
  Arms: Second-line therapy alone

SUMMARY:
Patients with glioblastoma face a grim prognosis. Despite recent advancement in neurosurgical technology and neuro-oncology glioblastomas almost invariably progress or recur after a median of 4-8 months. The strategy to repeat tumor resection at recurrence in order to minimize tumor load and thus to facilitate subsequent second-line therapy has been shown to be feasible and safe.

However, evidence for a survival benefit of surgery for recurrent glioblastoma is scarce and relies entirely on retrospective analyses. While most retrospective analyses report an apparent survival benefit, an EORTC meta-analysis on second-line therapies found no survival difference in patients with or without surgery at recurrence. With regard to the risks and costs inherent to surgery for glioblastoma, a randomized controlled trial is required.

The purpose of the study is to compare the effect of craniotomy and tumor resection followed by adjuvant second-line therapy to no surgery followed by second-line therapy on overall survival, neurological status, and quality of life. Analysis of overall survival will be used to improve sample size estimation of a subsequent phase III trial for craniotomy and tumor resection of glioblastoma recurrence in cooperation with the EORTC.

DETAILED DESCRIPTION:
Background

Glioblastoma is a malignant, locally invasive brain tumor whose prognosis remains grim despite various intense treatment modalities. In the past, radical surgery was met with skepticism due to the aggressive infiltrative character of the tumor. However, an increasing number of retrospective studies over the last decade suggest a survival benefit for surgery. A recent post-hoc analysis of a randomized controlled trial on the use of the surgical adjunct 5-ALA reported a prolonged overall survival from 11.9 to 16.7 months (evidence level 2a) after more extensive resection. Thus, maximal safe resection has become a mainstay of treatment for newly diagnosed glioblastoma, followed by adjuvant radio-chemotherapy.

Glioblastoma almost invariably recurs after a median of 6.9 months, leaving but few options for further treatment. Recurrence of glioblastoma after surgery and concomitant adjuvant therapy represents an additional therapeutic challenge and may be treated with second-line pharmacotherapy. In addition, a second surgery may also be considered in highly selected patients.

The rationale for surgery - maximum safe resection - is to prolong survival through reduction of tumor load, and, maybe due to an increased efficacy of adjuvant treatment. However, surgery carries risks of complications, that may result in a decreased functional and survival outcome. The crucial question therefore is whether, to what extent, and at what costs in terms of neurological risks a second resection prolongs survival.

Objective

The primary objective of this randomized trial is to compare survival outcome after surgery followed by adjuvant second-line therapy to no surgery followed by second-line therapy in recurrent glioblastoma. An auxiliary objective to primary objective is to compare the survival outcomes of operated patients to control in the subgroups stratified by extent of resection: incomplete resection (non-CRET) vs complete resection (CRET).

Secondary objectives are: assessment of recruitment for all screened patients, comparison of progression-free survival between treatment arms, evaluation of crossover and comparison of patient quality of life between treatment arms.

Safety objectives are: to assess neurological deficits, local infections and morbidity associated to surgery and hospital stay after surgery and during follow-up.

Methods

All patients (≥18 years) with a radiological suspicion of first recurrence of glioblastoma are screened for this trial. Patients eligible for study participation are informed on the treatment options for recurrent glioblastoma (surgery followed by adjuvant second-line therapy, second-line therapy, or palliative therapy alone) by the center investigators. Patients randomized to the control group will receive second-line therapy according to local guidelines. Patients randomized to the interventional group will receive a craniotomy and resection of the tumor followed by adjuvant second-line therapy. Outcome will be measured at 3 months intervals.

Recruitment rate and reason for non-inclusion will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ≥18 years of age
* Prior resection of glioblastoma confirmed by histology
* Glioblastoma pretreated with standard radiotherapy without or with temozolomide
* First progression according to RANO criteria
* First progression not within 3 months after completion of radiation therapy
* Complete removal of contrast-enhancing lesion considered feasible without significant risk of permanent speech or motor function according to MRI as confirmed by study eligibility committee after screening and prior to recruitment
* No encroachment of the M1 or A1 segments of the medial and anterior cerebral artery on MRI
* No contrast enhancement in presumed speech and primary motor areas on MRI
* No midline shift on MRI
* No contrast enhancing ventricular spread, multifocal recurrence, meningeosis carcinomatosa or infiltration of the contra-lateral hemisphere on MRI
* No contra-indication for surgery
* Good functional status (KPS ≥ 70)

Exclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-05-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival from the date of inclusion | From the date of inclusion until death/end of study, assessed up to 5.7 years

SECONDARY OUTCOMES:
Recruitment rate for all screened patients | Screening and inclusion
Progression-free survival | From the date of inclusion until the date of objective progression or the date of patient's death, whichever occurs first, assessed up to 5.7 years
Morbidity of surgery | Every 3 months up to 2 years or until death, assessed up to 5.7 years
Total number of days spent at home after recurrence | From the date of inclusion until death/end of study, assessed up to 5.7 years
Total number of days spent outside home after recurrence | From the date of inclusion until death/end of study, assessed up to 5.7 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Schucht, Prof. Dr. med., Principal Investigator — Dep. of Neurosurgery, Inselspital Bern
Locations (25):
- Austria (3):
  - Universitätsklinikum Innsbruck, Innsbruck
  - Johannes Kepler University Linz University, Clinic for Neurosurgery, Linz
  - Medical University of Vienna, Department of Neurosurgery, Vienna
- France (8):
  - Centre Hospitalier Universitaire Dijon Bourgogne, Department of Neurosurgery, Dijon
  - Hospices Civils de Lyon - CHU de Lyon, Department of Neuro-Oncology, Lyon
  - Assistance Publique - Hôpitaux de Marseille, Department of Neuro-Oncology, Marseille
  - Centre Hospitalier Universitaire de Nice, Department of Neurosurgery, Nice
  - Assistance Publique - Hôpitaux de Paris (AP-HP), Department of Neurosurgery, Paris
  - Centre Hospitalier Universitaire de Saint-Étienne, Department of Neurosurgery, Saint-Etienne
  - Institut de Cancérologie Strasbourg Europe (ICANS), Department of Oncology, Strasbourg
  - Centre Hospitalier Régional et Universitaire de Tours (CHRU Tours), Department of Neurosurgery, Tours
- Germany (2):
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Münster, Münster
- Department of Neurosurgery, Hospital of Larissa & General Hospital of Larissa, Larissa, Greece
- Netherlands (3):
  - Department of Neurosurgery, Amsterdam University Medical Center, Amsterdam
  - Department of Neurosurgery, Radboud University Medical Center, Nijmegen, Nijmegen
  - Department of Neurosurgery, Haaglanden Medical Center, The Hague, The Hague
- Department of Neurosurgery, Centro Hospitalar Universitário Lisboa Norte - Hospital de Santa Maria, Lisbon, Portugal
- Department of Neurosurgery, L'Hospitalet de Llobregat, Barcelona, Barcelona, Spain
- Sweden (2):
  - University of Gothenburg, Department of Clinical Neuroscience, Gothenburg
  - University Hospital of Umeå, Department of Diagnostics and Intervention, Umeå
- Switzerland (4):
  - Universitätsspital Basel, Basel
  - Dep. of Neurosurgery, Bern University Hospital, Bern
  - Dep. of Neurosurgery, Centre hospitalier universitaire vaudois, Lausanne
  - Ospedale Regionale di Lugano, Lugano